CLINICAL TRIAL: NCT01706536
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of the Efficacy and Safety of EP-101 (SUN101) in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease: GOLDEN-2 (Glycopyrrolate for Obstructive Lung Disease Via Electronic Nebulizer)
Brief Title: A Study of the Efficacy and Safety of EP-101 ( (SUN101) in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease
Acronym: GOLDEN-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP-101-04 (SUN101)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- EP-101 Placebo (Placebo Comparator): EP-101 Placebo AM + EP-101 Placebo PM
  Interventions: Drug: Placebo
- EP 101 12.5 mcg (Experimental): EP-101 12.5 mcg AM + EP-101 12.5 mcg PM
  Interventions: Drug: EP-101 12.5 mcg
- EP-101 25 mcg (Experimental): EP-101 25 mcg AM + EP-101 25 mcg PM
  Interventions: Drug: EP-101 25 mcg
- EP-101 50 mcg (Experimental): EP-101 50 mcg AM + EP-101 50 mcg PM
  Interventions: Drug: EP-101 50 mcg
- EP-101 100 mcg (Experimental): EP-101 100 mcg AM + EP-101 100 mcg PM
  Interventions: Drug: EP-101 100 mcg

INTERVENTIONS:
Drug: Placebo — EP-101 Placebo AM + EP-101 Placebo PM
  Other Names: SUN101
  Arms: EP-101 Placebo
Drug: EP-101 12.5 mcg — EP-101 12.5 mcg AM + EP-101 12.5 mcg PM
  Other Names: SUN101
  Arms: EP 101 12.5 mcg
Drug: EP-101 25 mcg — EP-101 25 mcg AM + EP-101 25 mcg PM
  Other Names: SUN101
  Arms: EP-101 25 mcg
Drug: EP-101 50 mcg — EP-101 50 mcg AM + EP-101 50 mcg PM
  Other Names: SUN101
  Arms: EP-101 50 mcg
Drug: EP-101 100 mcg — EP-101 100 mcg AM + EP-101 100 mcg PM
  Other Names: SUN101
  Arms: EP-101 100 mcg

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel arm study. The study population will consist of subjects, 35 to 75 years of age, with a diagnosis of moderate to severe COPD per Global Initiative for Chronic Obstructive Lung Disease guidelines.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel arm study. The study population will consist of subjects, 35 to 75 years of age, with a diagnosis of moderate to severe COPD per Global Initiative for Chronic Obstructive Lung Disease guidelines (GOLD, 2011). The primary analysis will compare each of the EP-101 (SUN101) dose groups to placebo with respect to the change from baseline in morning trough FEV1 on Day 29. Trough FEV1 is defined as the mean of the two FEV1 values obtained at 23 hours 30 minutes and 24 hours after Day 28 AM dose (ie, approximately 12 hours after the previous PM dose).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 35 through 75 years, inclusive.
* A clinical diagnosis of moderate to severe COPD according to GOLD guidelines (2011).
* Current smokers or ex-smokers with at least 10 pack-year smoking history (eg, at least 1 pack/day for 10 years, or equivalent).
* Post-bronchodilator (following inhalation of ipratropium bromide MDI) FEV1 ≥ 30% and ≤ 70% of predicted normal value during the Screening Period.
* Post-bronchodilator (following inhalation of ipratropium bromide MDI) FEV1/FVC ratio < 0.70 during the Screening Period.
* Post-bronchodilator (following inhalation of ipratropium bromide MDI) improvement in FEV1 ≥ 12% and ≥ 100 mL during the Screening Period.
* Ability to perform reproducible spirometry according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines (2005).
* Subject, if female ≤ 65 years of age and of child bearing potential, must have a negative serum pregnancy test at screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control:

  * a. An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following study participation.
  * b. Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study.
  * c. Abstinence.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Current evidence or recent history of any clinically significant and unstable disease (other than COPD) or abnormality in the opinion of the Investigator that would put the subject at risk or which would compromise the quality of the study data; including but not limited to cardiovascular disease, myocardial infarction, cardiac failure, uncontrolled hypertension, life-threatening arrhythmias, uncontrolled diabetes, neurologic or neuromuscular disease, liver disease, gastrointestinal disease or electrolyte abnormalities.
* Current evidence or history of clinically significant abnormal cardiac rhythm and/or conduction findings, including Holter monitoring results during the Screening Period.
* Concomitant pulmonary disease or primary diagnosis of asthma.
* History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin
* Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 6 weeks prior to the Screening Period.
* Use of daily oxygen therapy > 10 hours per day.
* Use of systemic steroids within 3 months prior to the Screening Period.
* Respiratory tract infection within 6 weeks prior to or during the Screening Period.
* History of tuberculosis, bronchiectasis or other non-specific pulmonary disease.
* History of urinary retention or bladder neck obstruction type symptoms.
* History of narrow-angle glaucoma.
* Prolonged QTc interval (> 450msec for males and > 470msec for females) during the Screening Period, or history of long QT syndrome.
* Recent history (previous 12 months) of excessive use or abuse of narcotic/illegal drugs.
* History of hypersensitivity or intolerance to β2-agonists or anticholinergics.
* Participation in another investigational drug study where drug was received within 30 days prior to the Screening Period.
* Female subject who is pregnant or lactating

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sunovion Respiratory Development
Locations (26):
- United States (26):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Pulmonary Associates, PA, Phoenix, Arizona
  - California Research Medical Group, Inc., Fullerton, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Integrated Research Group, Riverside, California
  - Capital Allergy & Respiratory Disease Center, Sacramento, California
  - Institute of HealthCare Assessment, Inc., San Diego, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Georgia Clinical Research, Austell, Georgia
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - Veritas Clinical Specialities, LTD, Topeka, Kansas
  - Minnesota Lung Center, Minneapolis, Minnesota
  - American Health Research, Charlotte, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Sunstone Medical Research LLC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Greenville Pharmaceutical Research, Inc, Greenville, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - CU Pharmacuetical Research, Union, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia

REFERENCES:
- [Result] Donohue JF, Goodin T, Tosiello R, Wheeler A. Dose selection for glycopyrrolate/eFlow(R) phase III clinical studies: results from GOLDEN (Glycopyrrolate for Obstructive Lung Disease via Electronic Nebulizer) phase II dose-finding studies. Respir Res. 2017 Dec 4;18(1):202. doi: 10.1186/s12931-017-0681-z. PMID 29202767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 302 subjects, 294 completed the run-in period. 12 out of 294 subjects completed the run-in period, but did not enter the double-blind period. Total of 282 subjects entered the double-blind period.
  Specific details are outlined in the table below.
Groups:
- Placebo: Placebo AM + Placebo PM
  Placebo:AM +Placebo PM
Period: Overall Study
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Started | 57 | 55 | 54 | 57 | 59
Completed | 53 | 51 | 49 | 53 | 57
Not Completed | 4 | 4 | 5 | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 4 | 3 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1 | 0
Not completed — non compliance | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg | Total
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 36 | 40 | 36 | 42 | 184
  >=65 years | 27 | 19 | 14 | 21 | 17 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.29) | 60.9 (7.79) | 59.6 (8.98) | 59.4 (8.70) | 59.4 (7.65) | 60.5 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 30 | 24 | 34 | 147
  Male | 26 | 27 | 24 | 33 | 25 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 0 | 4
  Not Hispanic or Latino | 56 | 55 | 52 | 56 | 59 | 278
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 3 | 3 | 10 | 27
  White | 49 | 51 | 50 | 53 | 49 | 252
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 55 | 54 | 57 | 59 | 282

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Trough Forced Expiratory Volume in 1 Second (FEV1)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. Trough FEV1 was defined as the mean of the spirometry values collected at 23 hours 30 minutes and 24 hours after the in-clinic morning dose (i.e. approximately 12 hrs after the previous evening dose).
Time Frame: Baseline and Day 29
Population: The ITT population consisted of all subjects who were randomized to treatment and received at least 1 dose of double-blind study medication.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
liters | 0.0009 (0.16664) | 0.1055 (0.18013) | 0.1333 (0.26526) | 0.1336 (0.23813) | 0.1794 (0.21678)
Statistical Analysis 1: Comparison: Placebo vs EP 101 12.5 mcg; A sample size of 45 subjects per treatment arm provides approximately 80% power to detect a 0.12 L treatment difference in mean change in trough FEV1 between an active arm and the placebo arm at a significance level of 0.05 using a 2-group t-test and assumes a standard deviation for change in trough FEV1 of 200. Assuming a 20% discontinuation rate, approximately 55 subjects were enrolled into each treatment arm; Test type: Superiority; p = 0.0043, Least squares mean (SE); In order to control for Type I error rate, a gate keeping methodology was used; Least Squares Mean (SE) = 0.1168, 95% CI 2-sided [0.0369 to 0.1966], Standard Error of Mean 0.04055
Statistical Analysis 2: Comparison: Placebo vs EP-101 25 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0019, Least squares mean (SE) — In order to control for Type I error rate, a gate keeping methodology was used; Least Squares Mean (SE) = 0.1284, 95% CI 2-sided [0.0479 to 0.2089], Standard Error of Mean 0.04089
Statistical Analysis 3: Comparison: Placebo vs EP-101 50 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0004, Least squares mean (SE) — in order to control for Type 1 error rate, a gate keeping methodology was used; Least Squares Mean (SE) = 0.1462, 95% CI 2-sided [0.0667 to 0.2257], Standard Error of Mean 0.04037
Statistical Analysis 4: Comparison: EP-101 100 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Least squares mean (SE) — in order to control for type I error rate, a gate keeping methodology was used; Least Squares Mean (SE) = 0.1770, 95% CI 2-sided [0.0992 to 0.2548], Standard Error of Mean 0.03953

2. Secondary Outcome: The Standardized Change From Baseline FEV1 AUC(0-12)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Placebo: Placebo AM + Placebo PM
  Placebo AM + Placebo PM
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 5 | 57 | 59
liters | 0.0055 (0.15426) | 0.1370 (0.17082) | 0.1720 (0.24720) | 0.1066 (0.20512) | 0.1815 (0.18544)

3. Secondary Outcome: The Standardized Change From Baseline FEV1 AUC(12-24)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
Time Frame: Day 28
Population: A substudy of subjects in the ITT population consisted of subjects who were randomized to treatment and received at least 1 dose of double-blind study medication and who had extended spirometry measurements.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 24 | 26 | 24 | 25 | 26
liters | -0.0725 (0.16509) | 0.0578 (0.14054) | 0.0563 (0.27985) | 0.0692 (0.19252) | 0.1284 (0.21688)

4. Secondary Outcome: The Peak FEV1 Change From Baseline
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. Peak FEV1 is defined as the highest postdose FEV1 value within 4 hrs after the morning dose.
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 55 | 54 | 54 | 57 | 59
liters | 0.0931 (0.17808) | 0.2613 (0.18782) | 002960 (.0026303) | 0.2552 (0.22395) | 0.3165 (0.21409)

5. Secondary Outcome: The Number of Subjects With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events were those which first occurred or increased in severity or relationship to study drug after the first dose of double-blind study drug.
Time Frame: Baseline up to Day 28
Population: The safety population consisted of all subjects who were randomized to treatment and received at least 1 dose of double-blind study medication. Safety analyses were performed using the actual drug a subject received.
Measure: Number; unit: participants
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
participants | 15 | 19 | 18 | 18 | 17

6. Secondary Outcome: The Number of Subjects With Treatment-emergent Serious Adverse Events
Description: Treatment-emergent serious adverse events were those which first occurred or increased in severity or relationship to study drug after the first dose of double-blind study drug.
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
participants | 2 | 2 | 2 | 1 | 3

7. Secondary Outcome: The Number of Subjects With Treatment-emergent Adverse Events Leading to Study Medication Discontinuation
Description: as for outcome 5
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
participants | 2 | 3 | 4 | 3 | 1

8. Secondary Outcome: The Percentage of Subjects With Treatment-emergent Adverse Events
Description: as for outcome 5
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
percentage of participants | 26.3 | 34.5 | 33.3 | 31.6 | 28.8

9. Secondary Outcome: The Percentage of Subjects With Treatment-emergent Serious Adverse Events
Description: as for outcome 6
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
percentage of participants | 3.5 | 3.6 | 3.7 | 1.8 | 5.1

10. Secondary Outcome: The Percentage of Subjects With Treatment-emergent Adverse Events Leading to Study Medication Discontinuation
Description: as for outcome 5
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Number analyzed (Participants) | 57 | 55 | 54 | 57 | 59
percentage of participants | 3.5 | 5.5 | 7.4 | 5.3 | 1.7

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: SAEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment
Arm/Group | Placebo | EP 101 12.5 mcg | EP-101 25 mcg | EP-101 50 mcg | EP-101 100 mcg
Serious Adverse Events (participants affected / at risk) | 1/57 | 2/55 | 2/54 | 0/57 | 1/59
Other Adverse Events (participants affected / at risk) | 3/57 | 2/55 | 5/54 | 3/57 | 6/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | EP 101 12.5 mcg (N=55) | EP-101 25 mcg (N=54) | EP-101 50 mcg (N=57) | EP-101 100 mcg (N=59)
pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | EP 101 12.5 mcg (N=55) | EP-101 25 mcg (N=54) | EP-101 50 mcg (N=57) | EP-101 100 mcg (N=59)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following the completion of the study at all sites, Institution and Investigator shall be free to publish.